CLINICAL TRIAL: NCT03761563
Title: Clinical Evaluation of Fortilink® TETRAfuse® Interbody Fusion Device in Subjects With Degenerative Disc Disease (FORTE)
Brief Title: Clinical Evaluation of Fortilink® TETRAfuse® Interbody Fusion Device in Subjects With Degenerative Disc Disease
Acronym: FORTE
Status: Completed | Type: Observational
Sponsor: Xtant Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 1105 CL
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fortilink IBF System with TETRAfuse Technology — Cervical and lumbar fusion

SUMMARY:
This is a prospective, multi-center, non-randomized post-market evaluation designed to collect and evaluate data on the safety and performance of the Fortilink IBF System with TETRAfuse 3D Technology.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized post-market evaluation designed to collect and evaluate data on the safety and performance of the Fortilink IBF System with TETRAfuse 3D Technology.

There will be 3 arms in the study, one for each configuration of the Fortilink IBF system (Fortilink-C, Fortilink-TS and Fortilink-L). Up to 50 subjects will be enrolled in each study arm for a total of up to 150 subjects at up to 20 sites in the United States (US) and European Union (EU).

ELIGIBILITY:
Inclusion Criteria:

* The subject is skeletally mature and at least 18 years of age.
* The subject has degenerative disc disease (DDD) of the cervical spine with accompanying radicular symptom at one or two contiguous levels (Fortilink-C), or the subject has DDD and ≤ Grade 1 spondylolisthesis of the lumbar spine at one or two contiguous levels (Fortilink-TS and Fortilink-L).
* Subject plans to undergo one of the following procedures:

An anterior cervical interbody fusion at one to two continuous levels from C2-C3 to C7-T1 using autogenous or allogenic bone graft and supplemental fixation cleared and indicated for use at the proposed treatment level(s) (Fortilink-C), or

An interbody fusion in the lumbar spine at one to two continuous levels from L1-L2 to L5-S1 using autogenous or allogenic bone graft and supplemental fixation cleared and indicated for use at the proposed treatment level(s) (Fortilink-TS and Fortilink-L).

* The subject has undergone non-operative treatment of at least six weeks (Fortilink-C) or at least six months (Fortilink-TS and Fortilink-L) prior to treatment with the IBF system.
* The subject is willing and able to provide informed consent.
* The subject is willing and able to attend the protocol required follow-up visits and examinations.

Exclusion Criteria:

* The subject has an active infection
* The subject has had prior fusion attempt(s) or is undergoing revision of a previously implanted system at the involved level(s).
* The subject is a worker's compensation case, in active litigation related to the procedure or is a prisoner or ward of the state.
* The subject meets one or more of the contraindications outlined in the IFU.
* The subject is pregnant, nursing, or is planning to become pregnant in the next year.
* The subject has documented evidence of current substance abuse.
* The subject has other concurrent medical condition that, in the opinion of the investigator, does not make the subject a good candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects in this study will be candidates who undergo interbody fusion of hte spine due to degenerative disc disease using the Fortilink IBF device.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of cervical fusion evaluated by radiographic evidence | 12 months
Rate of lumbar fusion evaluated by radiographic evidence | 24 months

SECONDARY OUTCOMES:
Change in pain from baseline evaluated by use of subject-reported 100mm Visual Analogue Scale (VAS) | 1 month, 3 months, 6 months, 12 months, and 24 months
  The VAS pain scale ranges from 0 to 100 where 0 represents No Pain and 100 represents Unbearable Pain.
Radiographic findings by CT evaluation | 12 months and 24 months
Time to return to work | up to 24 months
Incidence of serious device related adverse events | up to 24 months
Incidence of serious procedure related adverse events | up to 24 months
Change in functional ability determined by Neck Disability Index (NDI) or Oswestry Disability Index (ODI) | 3 months, 6 months, 12 months, and 24 months
  The NDI is a subject questionnaire designed to assess neck pain and will only be completed by subjects who undergo cervical implants. The ODI is a subject questionnaire designed to assess back pain and will only be completed by subjects who undergo lumbar implants. Each questionnaire consists of a total score ranging from 0 to 100 where a lower score represents a better outcome and a higher score represents a worse outcome.
Change in quality of life determined by SF-12 questionnaire | 3 months, 6 months, 12 months, and 24 months
  SF-12 questionnaires scores are computed and range from 0 to 100 where a 0 score indicates the lowest level of health and 100 indicates the highest level of health.
Change in pain medication usage from baseline | 1 month, 3 months, 6 months, 12 months, and 24 months

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Los Angeles Orthopedic Institute, Sherman Oaks, California
  - Rocky Mountain Spine Clinic, Lone Tree, Colorado
  - Florida Back Institute, Boca Raton, Florida
  - South Florida Spine & Orthopaedics, Coconut Creek, Florida
  - Spine Institute of South Florida, Delray Beach, Florida
  - Indiana Spine Center, Indianapolis, Indiana
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - OrthoBethesda, Bethesda, Maryland
  - ReVive Spine Center, Niagara Falls, New York
  - The Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Spine MD, North Richland Hills, Texas
  - Northwood Ortho-Spine, The Woodlands, Texas